CLINICAL TRIAL: NCT05646667
Title: Interscalene Block Alone Versus Interscalene Block With Erector Spinae Plane Block for Shoulder Arthroscopy Anesthesia: A Randomized Controlled Trial
Brief Title: Interscalene Block Alone Versus Interscalene Block With Erector Spinae Plane Block for Shoulder Arthroscopy Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Islam Morsy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35915/10/22
Record Dates: First submitted 2022-12-04; First posted 2022-12-12 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Interscalene Block; Erector Spinae Plane Block; Shoulder Arthroscopy Anesthesia; Randomized Controlled Trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene with erector spinae plane block group (Experimental): Patients will receive interscalene brachial plexus block using 10 ml of bupivacaine 0.5% and ultrasound guided erector spinae plane block at thoracic (T2) using 10 ml of bupivacaine 0.5%.
  Interventions: Other: interscalene with Erector spinae plane block group
- Interscalene group (Experimental): Patients will receive interscalene brachial plexus block using 15 ml of bupivacaine 0.5%.
  Interventions: Other: Interscalene group

INTERVENTIONS:
Other: interscalene with Erector spinae plane block group — patients will receive interscalene brachial plexus block using 10 ml of bupivacaine 0.5% and US guided Erector spinae plane block at T2 using 10 ml of bupivacaine 0.5%.
  Arms: Interscalene with erector spinae plane block group
Other: Interscalene group — patients will receive interscalene brachial plexus block using 15 ml of bupivacaine 0.5%.
  Arms: Interscalene group

SUMMARY:
The aim of this study is to compare the effectiveness of interscalene brachial plexus block alone versus interscalene brachial plexus block +Erector spinae plane block in anesthesia for shoulder arthroscopy.

DETAILED DESCRIPTION:
Regional anesthetic techniques can control pain effectively, both at rest and on movement, allowing earlier mobilization without the adverse effects of opioids . Among the various types of regional anesthetic techniques, the interscalene brachial plexus block is a gold standard used nerve block technique for postoperative analgesia in patients undergoing shoulder surgery, as it has consistently been shown to significantly control.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Both genders,
* BMI < 40 kg/m2
* American Society of Anesthesiologists (ASA) physical status I-II
* Scheduled for elective shoulder arthroscopy.

Exclusion Criteria:

* Known allergy to local anesthetics,
* allergy to all opioid medications, diagnostic shoulder arthroscopic procedures,
* patients with chronic opioids,
* patients who converted to general anesthesia use and coagulopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Intraoperative fentanyl consumption | Intraoperative up to 4 hours
  If the patient complains of pain during surgery, fentanyl will be administered 1 µg/kg IV increments.

SECONDARY OUTCOMES:
Amount of 24hrs postoperative rescue analgesic consumption | 24 hours postoperatively
  Intravenous meperidine (0.5 mg/kg) will be administered if numerical pain rating scale (NRS) score of more than 3.
Degree of pain by Numerical pain rating scale | 24 hours postoperatively
  Postoperative pain (using NRS at admission) will be measured at PACU, 1h, 2hr. 4hr, 6hr, 8hr, 12hr, 18hr, and 24hrs postoperative. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable").
Time to first request of rescue analgesia. | 24 hours postoperatively
  Rescue analgesia in the form of IV meperidine (0.5 mg/kg) boluses if NRS >3. Time to the 1st rescue analgesic request will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Islam Morsy, MD, Principal Investigator — Tanta University
Locations (1):
- Islam Morsy, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the data will be available upon reasonable request from the principle investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: from one year after completion of the study.